CLINICAL TRIAL: NCT01980511
Title: Detection and Neurological Impact of CerebroVascular Events In Noncardiac Surgery PatIents: A COhort EvaluatioN
Acronym: NeuroVISION
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Health and Medical Research Fund (Other Government); Prince of Wales Hospital, Shatin, Hong Kong (Other); Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: NeuroVISION v4.0
Record Dates: First submitted 2013-09-19; First posted 2013-11-11 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Covert Postoperative Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The NeuroVISION Study will characterize the incidence, impact, and risk factors of covert stroke in adults undergoing noncardiac surgery. We will determine the incidence of acute covert stroke using an MRI study of the brain in the days following noncardiac surgery. We will characterize the epidemiology and the impact of covert stroke in patients undergoing noncardiac surgery, and its association with cerebral deoxygenation.

DETAILED DESCRIPTION:
At the University of Wisconsin a planned sub study of NeuroVISION is being conducted aiming to enroll 100 patients with additional cognitive testing, MRI sequences and a preoperative MRI scan.

At Hamilton Juravinski Hospital, Hamilton General Hospital, Auckland City Hospital and Prince of Wales Hospital a planned sub study of NeuroVISION (PAFS - Perioperative Atrial Fibrillation and Postoperative Stroke) is being conducted aiming to enroll 400 participants. The purpose of this sub-study is to determine the prevalence of AF(Atrial Fibrillation) before surgery (i.e. "background" AF), as well of the incidence of AF after surgery using the Icentia CardioSTAT "patch-like" single lead heart rhythm monitor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years old
* An anticipated hospital stay of at least 2 days after elective noncardiac surgery that occurs under general or neuraxial anesthesia
* Written informed consent for potential participation prior to noncardiac surgery

Exclusion Criteria:

* Contraindication to MRI (e.g. implanted devices not safe for MRI studies, claustrophobia)
* Unable or unwilling to attend the follow-up appointments
* Documented history of dementia
* Residing in a nursing home
* Undergoing carotid artery surgery or intracranial surgery
* Unable to complete neurocognitive testing due to language, vision or hearing impairment
* Unable to communicate with the research staff due to language barriers
* Patients who do not undergo their research MRI study after surgery
* Patients who do not complete a baseline MoCA questionnaire
* Patients who suffer an acute overt clinical stroke after the index surgery, but before their research MR study
* Previously enrolled in the NeuroVISION Study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing elective non-cardiac surgery, ≥ 65 years old and an anticipated hospital stay of at least 2 days after elective noncardiac surgery that occurs under general or neuraxial anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 1116 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Postoperative cognitive dysfunction | 1 year
  Our primary objective is to characterize the impact of postoperative covert stroke on neurocognitive function 1 year after elective noncardiac surgery, as measured by a decrease of two or more points on the Montreal Cognitive Assessment (MoCA) scale from preoperative baseline test to the 1-year follow-up.

SECONDARY OUTCOMES:
Incidence of acute postoperative covert stroke | 30 days
  We will detect acute postoperative covert stroke using an MR study of the brain that will be performed between postoperative days 2 and 9.
Clinical 30-day outcomes (rated yes/no) | 30 days
  Overt stroke, transient ischemic attack, death, myocardial infarction, myocardial injury after noncardiac surgery, nonfatal cardiac arrest, major adverse cardiovascular events, cardiac revascularization procedures, bleeding, new atrial fibrillation, hypotension, congestive heart failure, new acute renal failure, infection and sepsis
Clinical 1-year outcomes (rated yes/no) | 1 year
  Overt stroke, transient ischemic attack, death, myocardial infarction, nonfatal cardiac arrest, major adverse cardiovascular events (composite), congestive heart failure, new acute renal failure, dementia and mild cognitive impairment
Postoperative delirium | 30 days
  Delirium will be measured using the Cognitive Assessment Method (CAM).
Physical function after surgery as assessed using the Modified Rankin Scale | 30 days and 1 year
  Physical function will be measured using the Modified Rankin Scale. The Modified Rankin Scale is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people. The scale runs from 0-6, running from perfect health without symptoms to death. A higher score is worse.
Physical function after surgery as assessed using the Lawton Instrumental Activities of Daily Living (iADL) Scale | 30 days and 1 year
  Physical function will be measured using the Lawton Instrumental Activities of Daily Living (iADL) Scale. The Lawton Instrumental Activities of Daily Living Scale refers to people's daily self-care activities. It consists of 8 activities. A lower score is worse.
Quality of life after surgery | 30 days and 1 year
  We will use the EQ-5D questionnaire to assess the patients' health-related quality of life. EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life. The first part contains the EQ-5D descriptive system, comprising of 5 questions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. A higher score is worse. The second part is a vertical, visual analogue scale with the end-points of "best imaginable health state" and "worst imaginable health state". Scale runs from 0 to 100. A lower score is worse.
Depressive symptoms after surgery | 30 days and 1 year
  We will use the 5-question version of the Geriatric Depression Scale (GDS-5) to measure depressive symptoms. The 5-question version of the Geriatric Depression Scale scoring will be from 0 to 5. The higher values indicate increasing depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: P.J. Devereaux, MD, PhD, Principal Investigator — Population Health Research Institute; Marko Mrkobrada, MD, FRCPC, Principal Investigator — University of Western Ontario, Canada
Locations (11):
- University of Wisconsin, Madison, Wisconsin, United States
- Canada (3):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - University Hospital, London Health Sciences, London, Ontario
- Clinica Santa Maria, Providencia, Santiago Metropolitan, Chile
- Prince of Wales Hospital, Shatin, SAR, Hong Kong
- Narayana Health, Bangalore, India
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Auckland City Hospital, Auckland, New Zealand
- Hospital Cayetano Heredia, Lima, Peru
- Szpital Specjalistycznym, Krakow, Poland

REFERENCES:
- [Derived] Taylor NL, Wehrman J, Banks MI, Nair V, Pearce RA, Kunkel D, Shine JM, Prabhakaran V, Lennertz R, Sanders RD. Dysfunctional resting state network connectivity predicts postoperative delirium after major surgery. Br J Anaesth. 2025 Dec 30:S0007-0912(25)00844-X. doi: 10.1016/j.bja.2025.11.036. Online ahead of print. PMID 41475933
- [Derived] Taylor J, Wu JG, Kunkel D, Parker M, Rivera C, Casey C, Naismith S, Teixeira-Pinto A, Maze M, Pearce RA, Lennertz R, Sanders RD. Resolution of elevated interleukin-6 after surgery is associated with return of normal cognitive function. Br J Anaesth. 2023 Oct;131(4):694-704. doi: 10.1016/j.bja.2023.05.023. Epub 2023 Jun 27. PMID 37385855
- [Derived] Payne T, Taylor J, Casey C, Kunkel D, Parker M, Blennow K, Zetterberg H, Pearce RA, Lennertz RC, Sanders RD. Prospective analysis of plasma amyloid beta and postoperative delirium in the Interventions for Postoperative Delirium: Biomarker-3 study. Br J Anaesth. 2023 May;130(5):546-556. doi: 10.1016/j.bja.2023.01.020. Epub 2023 Feb 25. PMID 36842841
- [Derived] Taylor J, Payne T, Casey C, Kunkel D, Parker M, Rivera C, Zetterberg H, Blennow K, Pearce RA, Lennertz RC, McCulloch T, Gaskell A, Sanders RD. Sevoflurane dose and postoperative delirium: a prospective cohort analysis. Br J Anaesth. 2023 Feb;130(2):e289-e297. doi: 10.1016/j.bja.2022.08.022. Epub 2022 Oct 1. PMID 36192219
- [Derived] Taylor J, Parker M, Casey CP, Tanabe S, Kunkel D, Rivera C, Zetterberg H, Blennow K, Pearce RA, Lennertz RC, Sanders RD. Postoperative delirium and changes in the blood-brain barrier, neuroinflammation, and cerebrospinal fluid lactate: a prospective cohort study. Br J Anaesth. 2022 Aug;129(2):219-230. doi: 10.1016/j.bja.2022.01.005. Epub 2022 Feb 8. PMID 35144802
- [Derived] Mrkobrada M, Chan MTV, Cowan D, Spence J, Campbell D, Wang CY, Torres D, Malaga G, Sanders RD, Brown C, Sigamani A, Szczeklik W, Dmytriw AA, Agid R, Smith EE, Hill MD, Sharma M, Sharma M, Tsai S, Mensinkai A, Sahlas DJ, Guyatt G, Pettit S, Copland I, Wu WKK, Yu SCH, Gin T, Loh PS, Ramli N, Siow YL, Short TG, Waymouth E, Kumar J, Dasgupta M, Murkin JM, Fuentes M, Ortiz-Soriano V, Lindroth H, Simpson S, Sessler D, Devereaux PJ. Rationale and design for the detection and neurological impact of cerebrovascular events in non-cardiac surgery patients cohort evaluation (NeuroVISION) study: a prospective international cohort study. BMJ Open. 2018 Jul 6;8(7):e021521. doi: 10.1136/bmjopen-2018-021521. PMID 29982215